CLINICAL TRIAL: NCT05125133
Title: A Household Randomized Control Trial of Insecticide-treated Eave Nets and Window Screens for Malaria Control in Chalinze District, Tanzania.
Brief Title: Evaluation of Insecticide-treated Eave Nets and Window Screens for Malaria Control in Tanzania.
Acronym: ITENs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ifakara Health Institute (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Swiss Tropical & Public Health Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ITENs
Record Dates: First submitted 2021-10-26; First posted 2021-11-18 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Malaria,Falciparum
Keywords: Insecticide-treated nets, Eaves, windows, Malaria, Tanzania.
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Intervention Model Description: Households allocated into Two arms to receive ITENs+ITWS installed or none with a 1:1 ratio at sub-village level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ITENs + ITWS (Experimental): Deltamethrin at 3g AI/kg, which corresponds to 144 mg/m², and PBO synergist at 10g/kg which corresponds to 480 mg/m² are coated in ITENs and ITWS nets that will be installed to cover opened eaves and windows. This was manufactured by Moon Netting FZCO, United Arab Emirates.
  Interventions: Other: ITENs + ITWS
- Negative arm (No Intervention): The houses allocated NOT to receive ITENs and ITWS.

INTERVENTIONS:
Other: ITENs + ITWS — A dual active ingredient (dual AI) Insecticide-Treated Eave nets (ITENs) in combination with Insecticide Treated Window screens (ITWS) for house modification.
  Arms: ITENs + ITWS

SUMMARY:
This is a household randomized trial of a new tool for house modification, Insecticide-Treated Eave nets (ITENs) in combination with insecticide-treated window screens (ITWS), coated with a dual active ingredient (dual AI): Deltamethrin at 3g AI/kg, which corresponds to 144 mg/m² and PBO synergist at 10g/kg which corresponds to 480 mg/m², as used in the so-called dual-AI LLIN or "resistance breaking" nets for resistance malaria vector control.

Four hundred and fifty (450) households with intact walls, opened eaves, and those without screens or nets on the windows in Chalinze district, Tanzania will be eligible and only recruited upon written informed consent. The households will be randomly allocated into two arms: one with ITENs and ITWS installed and the other without.

The primary outcome will be malaria parasite detection in household residents aged over 6 months old using a quantitative Polymerase Chain Reaction (qPCR) at approximately 12 months post-installation, coinciding with the long rainy season.

DETAILED DESCRIPTION:
In Tanzania, long-lasting insecticidal nets (LLINs) contributed to the high reduction of malaria in the last decade. However, malaria reduction in Tanzania is threatened due to increasing insecticidal resistance of malaria vectors, low access to LLIN, LLINs not lasting up to three years, and net usage compliance. Therefore, it is evident that an additional cost-effective vector control tool is required that may confer protection against resistant malaria vectors, protect every member of the household, requires little or less compliance to use after distribution, and lasts longer.

The proposed additional vector control tool for trial is the Insecticide-Treated Eave nets (ITENs) in combination with Insecticide Treated Window screens (ITWS) for house modification. The tool is coated with a dual active ingredient (dual AI): Deltamethrin at 3g AI/kg, which corresponds to 144 mg/m², and PBO synergist at 10g/kg which corresponds to 480 mg/m², which are coated at the same concentration in insecticide-treated nets that are already in use in the population to control pyrethroid-resistant mosquitoes. These can protect everyone in the house by blocking mosquito entry and killing mosquitos that contact them to protect everyone in the community.

In this trial, 450 households will be randomly allocated into two arms. One arm with ITENs & ITWS installed and the other without to serve as the control arm. The 450 households are recruited and assigned codes during baseline data collection. The assigned codes are randomized to either of the two arms by simple randomization in STATA and stratified by sub-village.

Approximately 6 months and 12 months post-installation, coinciding with the rainy seasons, clinical officers will screen for malaria parasites in household residents of over 6 months old (it is estimated that 4.4 persons reside in each household, thus approx. 1,800 persons will be screened for malaria per survey) in both arms and confirmation of malaria parasite will be done using qPCR analysis as the primary assessment of the primary outcome. As a point of care, SD Bioline Malaria Ag Pf/Pan rapid diagnostic test (RDT) as per Tanzanian guidelines will also be conducted on all household residents. Any participant (s) with an axillary temperature of 37.5 degrees (fever) and that test positive using mRDT will be considered as a clinical malaria case. All malaria-positive participants will be treated using free Artemether Lumefantrine (ALu). This drug is approved by the national guideline for the treatment of uncomplicated malaria.

Other secondary objectives are:

* To evaluate malaria prevalence in households with ITENs & ITWS and those without at approximately 6 months post-installation, coinciding with the short rainy season.
* To determine the prevalence of clinical malaria defined by an axillary temperature of 37.5 degrees and above (fever) and mRDT malaria positive cases at approximately 6 months and 12 months post-installation, coinciding with the rainy seasons.
* To investigate the effect of ITENs and ITWS on the density of malaria vectors and nuisance (Culex quinquefasciatus) mosquitoes in the community at approximately 6 months and 12 months post-installation, coinciding with the rainy seasons using Centres for Disease Control (CDC) light traps.
* To assess the number of fabric in meters and time of installing the intervention (feasibility of scaling-up ITENs and ITWS use) in local houses in the field during installation.
* To assess the adverse effects of ITENs and ITWS in the community.
* To determine the attrition and fabric integrity of ITENs and ITWS in the field post 6 months and 12 months of installation.
* To determine the mortality induced by (bioefficacy) ITENs and ITWS on laboratory-reared mosquitoes post 12 months of installation.
* To determine the insecticide retainment of ITENs and ITWS post 12 months of installation.
* To assess the acceptability of ITENs and ITWS to the local community post 6 months and 12 months of installation.

ELIGIBILITY:
Inclusion Criteria:

* Residents of study households' members.

Exclusion Criteria:

* None residence.
* Pregnant women.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Plasmodium falciparum parasite. | Approximately 12 months post-installation, coinciding with the long rainy season.
  Prevalence of plasmodium falciparum parasite measured by qPCR among residents over 6 months old in houses with ITENs & ITWS compared to houses without.

SECONDARY OUTCOMES:
Prevalence of Plasmodium falciparum parasite. | Approximately 6 months post-installation, coinciding with the short rainy season.
  Prevalence of plasmodium falciparum parasite in households' residents of over 6 months old with ITENs & ITWS compared to those without using qPCR analysis.
Clinical malaria. | Approximately 6 months and 12 months post-installation, coinciding with the rainy seasons.
  The prevalence of clinical malaria cases defined by an axillary temperature of 37.5 degrees (fever) and positive mRDT in houses with ITENs and ITWS compared to the houses without.
The density of malaria vectors and nuisance mosquitoes density. | Approximately 6 months and 12 months post-installation, coinciding with the rainy seasons.
  Indoor density of malaria vector and nuisance mosquitoes in houses with ITENs & ITWS compared to houses without measured using Centres for Disease Control (CDC) light traps.
ITENs & ITWS fabric cost | Baseline (During installation of ITENs & ITWS)
  The number of metres of material applied to houses.
ITENS & ITWS time duration | Baseline (During installation of ITENs & ITWS)
  Time in hours to install the intervention.
Adverse effects | Approximately one month post installation.
  The number of participants with perceived adverse effects from ITENs and ITWS.
Attrition | Appriximately 6 months and 12 months post installation.
  Determination of the physical presence of ITENs and ITWS in the field.
Fabric integrity | Appriximately 6 months and 12 months post installation.
  Determination of the number of holes in ITENs and ITWS in the field.
The induced mosquito mortality of ITENs and ITWs on the population of laboratory-reared mosquitoes. | Approximately 12 months post installation.
  The bioefficacy (% induced mosquito mortality) of ITENs and ITWS after field use through WHO bioassays.
Insecticide retainment | Appriximately 12 months post installation.
  The retention of deltamethrin and PBO in grams per kg will be assessed through high performance liquid chromatography.
Use of ITENs and ITWS | Approximately 6 months and 12 months post installation.
  Community opinions of ITENs and ITWS will be sought through questionnaires and Focus Group Discussions.

CONTACTS AND LOCATIONS:
Overall Officials: John Bradley, PhD, Study Director — London School of Hygiene and Tropical Medicine
Locations (1):
- Vector Control Product Testing Unit Facility, Bagamoyo, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Data will be disseminated by a report to the sponsor, followed by peer-reviewed publications targeted towards consumers, scientists, and policy-makers. We will publish the results and data sets in open-access, indexed, peer-reviewed journals, making the findings and the data publicly available to all stakeholders. Data obtained from the study will be presented at international conferences and stakeholder meetings including the National Malaria Control Program, with priority given to the young scientists to practice their presentation and collaboration skills. At the end of the project, a meeting will be held to update the local community and the District Medical Officer (DMO), to present findings and answer any questions arising.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available at the end of the trial once it is analysed and published.
Access Criteria: Peer-reviewed open-source journals.

REFERENCES:
- [Background] Gnanguenon V, Azondekon R, Oke-Agbo F, Beach R, Akogbeto M. Durability assessment results suggest a serviceable life of two, rather than three, years for the current long-lasting insecticidal (mosquito) net (LLIN) intervention in Benin. BMC Infect Dis. 2014 Feb 8;14:69. doi: 10.1186/1471-2334-14-69. PMID 24507444
- [Background] Matiya DJ, Philbert AB, Kidima W, Matowo JJ. Dynamics and monitoring of insecticide resistance in malaria vectors across mainland Tanzania from 1997 to 2017: a systematic review. Malar J. 2019 Mar 26;18(1):102. doi: 10.1186/s12936-019-2738-6. PMID 30914051
- [Background] Mboera LE, Mweya CN, Rumisha SF, Tungu PK, Stanley G, Makange MR, Misinzo G, De Nardo P, Vairo F, Oriyo NM. The Risk of Dengue Virus Transmission in Dar es Salaam, Tanzania during an Epidemic Period of 2014. PLoS Negl Trop Dis. 2016 Jan 26;10(1):e0004313. doi: 10.1371/journal.pntd.0004313. eCollection 2016 Jan. PMID 26812489
- [Background] Mboma ZM, Overgaard HJ, Moore S, Bradley J, Moore J, Massue DJ, Kramer K, Lines J, Lorenz LM. Mosquito net coverage in years between mass distributions: a case study of Tanzania, 2013. Malar J. 2018 Mar 1;17(1):100. doi: 10.1186/s12936-018-2247-z. PMID 29490649
- [Result] Gleave K, Lissenden N, Richardson M, Choi L, Ranson H. Piperonyl butoxide (PBO) combined with pyrethroids in insecticide-treated nets to prevent malaria in Africa. Cochrane Database Syst Rev. 2018 Nov 29;11(11):CD012776. doi: 10.1002/14651858.CD012776.pub2. PMID 30488945
- [Derived] Odufuwa OG, Moore SJ, Mboma ZM, Mwanga R, Matwewe F, Hofer LM, Matanila I, Abbasi S, Rashid MA, Philipo R, Kihwele F, Moore J, Nguyen H, Bosselmann R, Skovmand O, Stevenson JC, Muganga JB, Bradley J. A household randomized-control trial of insecticide-treated screening for malaria control in unimproved houses in Tanzania. Malar J. 2025 Jun 8;24(1):182. doi: 10.1186/s12936-025-05434-2. PMID 40484966

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT05125133/Prot_ICF_000.pdf